CLINICAL TRIAL: NCT00513097
Title: Curbing Tobacco Use in Suburban and Rural Schools
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2005-0914; NCI-2011-02826 (Registry Identifier: NCI CTRP); 2R01CA081934-05A1 (NIH)
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Tobacco Use Cessation
Keywords: Epidemiology; Cancer Prevention; Smoking Cessation; Smoking Prevention; Focus Groups
MeSH Terms: conditions — Tobacco Use Cessation; Smoking Cessation | interventions — Focus Groups; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Smoking Prevention & Cessation Program (Experimental)
  Interventions: Behavioral: Smoking Prevention Program; Behavioral: Focus Group; Behavioral: Survey

INTERVENTIONS:
Behavioral: Smoking Prevention Program — Interactive internet, computer-based activities (like games) with questions about thoughts on smoking and tobacco.
Behavioral: Focus Group — A total of 24 focus groups will be held relating to the topics of smoking prevention and cessation.
Behavioral: Survey — On-line evaluations and questionnaires

SUMMARY:
Primary, secondary, and tertiary specific aims are to answer the following questions about interactive, Internet-based tobacco control intervention directed towards 10th-graders:

1. Smoking Prevention (primary): Does the intervention result in a lower incidence of smoking initiation compared to standard care?
2. Smoking Cessation (primary): Does the intervention result in higher rates of smoking cessation compared to standard care?
3. Reduction of Spit Tobacco Use (secondary): Does the intervention have an impact on spit tobacco use compared to standard care?
4. Stages of Change (tertiary): Does the intervention have an impact on progression through the stages of smoking and spit tobacco acquisition and cessation compared to standard care?
5. Mediating Variables (tertiary): How are mediating variables associated with tobacco-use onset and cessation?
6. Testing Predictors: Investigate established and recently elucidated predictors of susceptibility to smoking at baseline and 12-month follow-up.
7. Develop/Validate Spit Tobacco Measures: Investigate predictors of susceptibility of spit tobacco use at baseline and 12-month follow-up
8. Testing Measures Across Race/Ethnicity: Explore predictors of susceptibility to smoking at baseline and 12-month follow-up to determine whether predictors differ among White, African-American, and Hispanic students.

DETAILED DESCRIPTION:
The proposed study will test the effectiveness of the Internet-based cigarette smoking and spit tobacco (ST) prevention and cessation in-class curriculum for rural teens. Supplemented by "cyber-support" (chat room and bulletin board), the intervention program also will make use of a human social support environment (via trained school personnel, chat rooms, bulletin boards). The study will use a nested cohort design in which high schools are the unit of design, allocation, and analysis. Tenth-grade students (ages 14-16) within each intervention school will receive a 7-week interactive, Internet-based tobacco prevention and cessation curriculum. Using computerized surveys, study participants will be evaluated at baseline, 6-month, 12-month, and 18-month follow-ups. The study has been designed to permit analyses sensitive enough to detect differences for the two primary hypotheses: reductions in smoking initiation and smoking cessation. Trends in ST use after exposure to the intervention program will also be assessed. The design will also permit analysis of stage-of-change dynamics and mediators for both acquisition and cessation of both forms of tobacco.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 14-16 years of age (9th and 10th-graders) who speak, read and write English
2. Subjects are students from schools located in suburban and rural communities approximately 200 miles from Houston.
3. Subjects with approved parental consent

Exclusion Criteria:

1) Disruptive individuals who are not able to work with the program

Ages: 14 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1289 (Actual)
Dates: Start 2006-07-25 (Actual); Primary Completion 2017-10-18 (Actual); Study Completion 2017-10-18 (Actual)

PRIMARY OUTCOMES:
Reductions in smoking initiation | Baseline, 6-month, 12-month, and 18-month

SECONDARY OUTCOMES:
Smoking cessation | Baseline, 6-month, 12-month, and 18-month

CONTACTS AND LOCATIONS:
Overall Officials: Alex Prokhorov, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org